CLINICAL TRIAL: NCT02409602
Title: Comparison of the Dorsal Clitoral Artery Doppler Examination Results and the Female Sexual Function Index in Women With Postpartum Hemorrhage Who Underwent Bilateral Internal Iliac Artery Ligation and Age-matched Healthy Postpartum Women
Brief Title: Influence of BIIAL Following PPH on Dorsal Clitoral Artery Blood Flow and FSFI
Status: Completed | Type: Observational
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Baris KAYA, Assistant Professor, MD, Near East University, Turkey
Other Study IDs: CLITDOP-001
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Bilateral Iliac Artery Ligation; Postpartum Hemorrhage
Keywords: Ultrasonography, Doppler, Color; Postpartum hemorrhage; Bilateral iliac artery ligation; Dorsal clitoral artery
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Women with BIIAL: Women who underwent bilateral internal iliac artery ligation due to postpartum hemorrhage within last 2 months
  Interventions: Other: Doppler ultrasonographic examination
- Healthy puerperal women: Age-matched healthy puerperal women who delivered within last 2 months
  Interventions: Other: Doppler ultrasonographic examination

INTERVENTIONS:
Other: Doppler ultrasonographic examination — Dorsal clitoral artery Doppler ultrasonographic examinations will be performed regularly in 3rd and 6th months after delivery, in order to evaluate the possible effects of BIIAL on clitoral blood flow.

SUMMARY:
Dorsal clitoral artery Doppler examinations in women with bilateral internal iliac artery ligation due to postpartum hemorrhage (study group) and age-matched healthy puerperal women were performed regularly in the postoperative period, in order to evaluate possible effects of BIIAL on clitoral blood flow.

DETAILED DESCRIPTION:
Women who underwent bilateral internal iliac artery ligation due to postpartum hemorrhage in Gaziantep Cengiz Gokcek Maternity Hospital, Gaziantep Turkey and Near East University, Department of Obstetrics and Gynecology, Mersin, Turkey comprise the study group. The control group consists of age-matched healthy women who delivered in last 2 months.

Dorsal clitoral artery Doppler examinations will be performed in both case and control groups regularly in the postoperative period in 3rd and 6th months, in order to evaluate the possible effects of BIIAL on clitoral blood flow. Ultrasound is performed using a Mindray DC-7 Ultrasound System (China) equipped with linear 7.5 MHz probe. Each woman was scanned in the gynecological position. The translabial probe is placed on the clitoris sagittally and transversely without applying any pressure force. After identifying the clitoral artery using colour flow mapping, the Doppler probe is positioned over the vessel and at least three sequential Doppler wave forms are obtained. The following parameters are analysed: peak systolic velocity (PSV), end diastolic velocity (EDV), resistive index (RI), pulsatile index (PI) and systolic/diastolic (S/D) ratio. The measurements are performed by the same radiologist.

Finally a Female Sexual Fantasy Questionnaire (FSFQ) is performed.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 year-old women who underwent bilateral internal iliac artery ligation (BIIAL) due to postpartum hemorrhage
* Age-matched healthy puerperal women

Exclusion Criteria:

* Known Diabetes Melitus or cardiovascular disease
* Known affection disorder before or during pregnancy
* B-lynch procedure, ligation of uterine or ovarian artery, hysterectomy and salphingooophorectomy following postpartum hemorrhage
* Known functional sexual disorder before pregnancy
* Postoperative endometritis or other puerperal infections
* Postoperative thromboembolic incidence
* Cessation of breastfeeding in puerperal period

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18-35 year old women with postpartum hemorrhage who did and did not undergo bilateral internal iliac artery ligation (BIIAL)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Peak systolic velocity (PSV) | 6 months
Peak diastolic velocity (PDV) | 6 months
Resistive index (RI) | 6 months
End diastolic velocity (EDV) | 6 Months
Pulsatile index (PI) | 6 months
Systolic/diastolic (S/D) ratio | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Near East University, Obstetrics and Gynecology, Mersin, Trnc, Turkey (Türkiye)

REFERENCES:
- [Derived] Kaya B, Usluogullari B, Yurttutan N, Sahan MH, Guralp O, Malik E. Does ligation of internal iliac artery for postpartum hemorrhage affect clitoral artery blood flow and postpartum sexual functions? Eur J Obstet Gynecol Reprod Biol. 2017 Dec;219:124-128. doi: 10.1016/j.ejogrb.2017.10.029. Epub 2017 Oct 31. PMID 29102811